CLINICAL TRIAL: NCT03101436
Title: Extra Virgin Olive Oil and Red Wine Polyphenols in the Modulation of Fecal Microbiota: an Interventional Study
Brief Title: Extra Virgin Olive Oil, Red Wine Polyphenols and Fecal Microbiota
Acronym: OLIWINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JCMI2017
Record Dates: First submitted 2017-03-29; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: Insulin Resistance; Extra Virgin Olive Oil; Red Wine; Diet; Microbiota
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Phase I: Intervention with Diet (Extra Virgin Olive Oil) Washout Period Phase I: Intervention with Diet (Red Wine)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lean Subjects (Experimental): Part 1: Mediterranean diet with added extra virgin olive oil (80 gr per day) (1 month)
  Washout 15 days
  Part 2: Mediterranean diet with added Red Wine (270 ml per day) (1 month)
  Interventions: Dietary Supplement: Extra Virgin Olive Oil and Red Wine
- Obese Subjects (Experimental): Part 1: Mediterranean diet with added extra virgin olive oil (80 gr per day) (1 month)
  Washout 15 days
  Part 2: Mediterranean diet with added Red Wine (270 ml per day) (1 month)
  Interventions: Dietary Supplement: Extra Virgin Olive Oil and Red Wine

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive Oil and Red Wine — Phase I: Extra VIrgin Olive Oil 80 grams per day (1 month)
  Washout Period: 15 days
  Phase II: Red Wine (270 ml per day) (1 month)

SUMMARY:
In this study, the investigators will evaluate the prebiotic effect of a moderate intake of extra virgin olive oil or red wine on the modulation of gut microbiota composition and the improvement of cardiometabolic factors in obese and lean adults subjects.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients (body mass index (BMI= or > 30kg/m2) with high insulin resistance (measured by Homeostasis Model Assessment Insulin Resistance Index (HOMA-IR) > 5.5.
* Lean subjects (BMI< 28kg/m2) with low insulin resistance (HOMA-IR< 3.3).

Exclusion Criteria (all patients):

* Type 2 diabetes
* Acute or chronic infection
* Inflammatory disease or endocrine disorders.
* History of cancer.
* Anti-inflammatory, corticosteroid, hormone, or antibiotic drug treatment
* A history of alcohol abuse or drug dependence
* A restrictive diet or a weight change ≥5 kg during the 3 months prior to the study.
* Intake of prebiotics, probiotics, vitamin supplements or any other medical treatment influencing intestinal microbiota during the 3 months before the start of the study or during the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2015-05-06 (Actual); Study Completion 2015-05-06 (Actual)

PRIMARY OUTCOMES:
Microbiota Changes | 1 month
  Changes in microbiome composition

SECONDARY OUTCOMES:
Trimethylamine N-oxide (TMAO) production | 1 month
  Modifications in Trimethylamine N-oxide (TMAO) production
Insulin Resistance | 1 Month
  Modifications in Insulin Resistance (measured by Homeostasis Model Assessment Insulin Resistance Index (HOMA-IR))
Lipid Profile | 1 Month
  Changes in lipid profile (LDL, HDL, total cholesterol, triglycerides)

IPD SHARING:
Plan to Share IPD: No